CLINICAL TRIAL: NCT06603376
Title: A Randomized, Multicenter, Controlled Study of Irinotecan Hydrochloride Liposome Injection (Ⅱ) Combined with Fluorouracil, Folinic Acid, Vermofenib and Cetuximab in First-line Treatment of BRAFV600E Mutated Advanced Colorectal Cancer
Brief Title: Irinotecan Hydrochloride Liposome Injection (Ⅱ) Combined with Fluorouracil, Folinic Acid, Vermofenib and Cetuximab in First-line Treatment of BRAFV600E Mutated Advanced Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Yuan-Sheng Zang, Professor, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMPROVEMENT-2
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Carcinoma
Keywords: colorectal cancer; BRAF V600E; chemotherpay; Vemurafenib; Cetuximab; irinotecan hydrochloride liposome injection
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Vemurafenib; Cetuximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FOLFIRI + Vemurafenib + Cetuximab (Experimental): Experimental Group: Liposomal Irinotecan Hydrochloride Injection (II): 60 mg/m², intravenous infusion over at least 90 minutes, on day 1; Leucovorin: 400 mg/m², intravenous infusion over 2 hours, on day 1; 5-FU: 400 mg/m², intravenous bolus; 5-FU: 2400 mg/m², continuous infusion over 46-48 hours, on day 1; Cetuximab: 500 mg/m², intravenous infusion over at least 2 hours, on day 1; Vemurafenib: 720 mg, orally twice daily. Repeat every 2 weeks.
  Interventions: Drug: FOLFIRI + Vemurafenib + Cetuximab
- FOLFIRI ± Bevacizumab (Active Comparator): Control Group: Liposomal Irinotecan Hydrochloride Injection (II): 60 mg/m², intravenous infusion over at least 90 minutes, on day 1; Leucovorin: 400 mg/m², intravenous infusion over 2 hours, on day 1; 5-FU: 400 mg/m², intravenous bolus; 5-FU: 2400 mg/m², continuous infusion over 46-48 hours, on day 1; Bevacizumab: 5 mg/kg, intravenous infusion, on day 1. Repeat every 2 weeks.
  Interventions: Drug: FOLFIRI ± Bevacizumab

INTERVENTIONS:
Drug: FOLFIRI + Vemurafenib + Cetuximab — Liposomal Irinotecan Hydrochloride Injection (II): 60 mg/m², intravenous infusion over at least 90 minutes, on day 1; Leucovorin: 400 mg/m², intravenous infusion over 2 hours, on day 1; 5-FU: 400 mg/m², intravenous bolus; 5-FU: 2400 mg/m², continuous infusion over 46-48 hours, on day 1; Cetuximab: 500 mg/m², intravenous infusion over at least 2 hours, on day 1; Vemurafenib: 720 mg, orally twice daily. Repeat every 2 weeks.
  Arms: FOLFIRI + Vemurafenib + Cetuximab
Drug: FOLFIRI ± Bevacizumab — Liposomal Irinotecan Hydrochloride Injection (II): 60 mg/m², intravenous infusion over at least 90 minutes, on day 1; Leucovorin: 400 mg/m², intravenous infusion over 2 hours, on day 1; 5-FU: 400 mg/m², intravenous bolus; 5-FU: 2400 mg/m², continuous infusion over 46-48 hours, on day 1; Bevacizumab: 5 mg/kg, intravenous infusion, on day 1. Repeat every 2 weeks.
  Arms: FOLFIRI ± Bevacizumab

SUMMARY:
Based on the upstream signaling features of BRAFV600E and the bypass feedback mechanisms, considering the pro-apoptotic effects of chemotherapy and the synergistic effects of targeted therapy, previous IMPROVEMENT trial creatively explored a balanced chemotherapy-targeted combination approach (FOLFIRI + Vemurafenib + Cetuximab) in advanced colorectal cancer patients with BRAF V600E mutaiton using a signle-arm study design, demonstrating significant therapeutic efficacy in these patietns . To further validate the effectiveness and safety of this regimen and to solidify its clinical value, it is crucial to conduct a randomized, controlled trial. Investigators plan to use the current standard regimen as a control to compare this strategy (FOLFIRI + Vemurafenib + Cetuximab) on a large cohort of patients with BRAFV600E-mutant advanced colorectal cancer in the first-line setting, focusing on its efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced colorectal adenocarcinoma confirmed by histology or cytology.
* Patients with BRAFV600E mutation confirmed by tissue or blood testing.
* Patients who have not received systemic therapy or who have experienced metastasis or recurrence 12 months after completing adjuvant therapy.
* Patients must have at least one measurable lesion according to RECIST 1.1 criteria.
* Patients who received local radiotherapy at least 3 weeks before the first drug treatment are allowed to enroll, but lesions evaluated by RECIST should not be within the radiation field.
* Patients aged ≥18 years and ≤80 years.
* ECOG performance status of 0-2.
* Expected survival of ≥12 weeks.
* Patients must have the ability to understand and voluntarily sign a written informed consent.
* Women of childbearing potential must have a negative pregnancy test within 7 days prior to the start of treatment. During the study, both the patient and their partner must use contraception.

Exclusion Criteria:

* Patients who have undergone major surgery or suffered severe trauma within 4 weeks prior to the first dose of the study drug.
* Patients with hypersensitivity to any component of the study regimen.
* Patients who are planning to conceive or are already pregnant.
* Patients with brain metastases who cannot accurately describe their condition.
* Patients with the following conditions within 6 months prior to the start of the study treatment: myocardial infarction, severe/unstable angina, congestive heart failure greater than NYHA Class 2, uncontrolled arrhythmias, etc.
* Abnormal laboratory test results:
* Absolute neutrophil count (ANC) <1,500/mm³;
* Platelet count <75,000/mm³;
* Total bilirubin >1.5 times the upper limit of normal (ULN); ALT (alanine aminotransferase) and AST (aspartate aminotransferase) >2.5 times ULN (for patients with liver metastasis >5 times ULN); Creatinine >1.5 times ULN;
* Patients who have had any cancer other than advanced colorectal cancer within five years prior to the start of the study treatment. Exceptions include cervical carcinoma in situ, cured basal cell carcinoma, and bladder epithelial tumors.
* Patients with a history of drug abuse, substance abuse, or alcohol dependence.
* Patients who are legally incapacitated or have limited civil capacity.
* Any other conditions deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Evaluation of tumor burden based on RECIST criteria through study completion, an average of 8 weeks
  Proportion of patients with reduction in tumor burden of a predefined amount, including complete remission and partial remission

SECONDARY OUTCOMES:
Progress Free Survival | Evaluation of tumor burden based on RECIST criteria until first documented progress or death through study completion, an average of 8 weeks
  Time from treatment beginning until disease progression or death from any cause
Overall Survival | From date of treatment beginning until the date of death from any cause, through study completion, an average of 8 weeks
  Time from treatment beginning until death from any cause
Deepness of response | Evaluation of tumor burden based on RECIST criteria through study completion, an average of 8 weeks
  Investigation of depth of response during first-line treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-Sheng Zang, Professor, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No